CLINICAL TRIAL: NCT05570786
Title: A Phase II, Randomized, Placebo-controlled, Double-blind, Multicenter Study to Investigate the Safety and Exploratory Efficacy of a Subdermal Implant-bioabsorbable Gestrinone Pellet for Pelvic Pain Secondary to Endometriosis Treatment
Brief Title: Subdermal Implant-bioabsorbable Gestrinone Pellet for Endometriosis Pelvic Pain Treatment
Acronym: GLADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Collaborators: Biós Farmacêutica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLADE
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Deep Endometriosis; Pelvic Pain
Keywords: Hormone Pellet Therapy; Implantable Hormone Pellets; Endometriosis; Pelvic pain
MeSH Terms: conditions — Pelvic Pain; Endometriosis | interventions — Gestrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gestrinone (Experimental): Subdermal implant-bioabsorbable gestrinone pellet (85 mg) All patients will undergo insertion of an intrauterine system of levonorgestrel release (Kyleena®) as a contraceptive method
  Interventions: Drug: Gestrinone
- Placebo (Placebo Comparator): Subdermal implant-bioabsorbable placebo pellet (cholesterol) All patients will undergo insertion of an intrauterine system of levonorgestrel release (Kyleena®) as a contraceptive method
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gestrinone — The intradermal gestrinone/placebo pellet will be inserted on the same day as the levonorgestrel intrauterine hormonal device (Kyleena®)
  Arms: Gestrinone
Drug: Placebo — Subdermal implant-bioabsorbable placebo pellet (cholesterol)
  Arms: Placebo

SUMMARY:
Pelvic pain is considered a symptom of multifactorial origin among which Endometriosis is the main gynecological cause affecting 5-10% of worldwide women in their reproductive years, negatively impacting their quality of life and work efficiency. Treatment of endometriosis-associated pelvic pain is challenging and there are surgical and/or hormonal treatments available with variable endpoints. Gestrinone is a synthetic derivative of 19-nortestosterone with anti-estrogen, anti-progestin, androgenic, and weak estrogen-like action. Previous studies show that the oral treatment with Gestrinone induced an improvement in symptoms associated with endometriosis but with adverse events such as androgenization and uterine bleeding. Parenteral administration of Gestrinone could be effective to treat pain symptoms secondary to endometriosis and minimize these adverse events. This study evaluates the safety and tolerability of subdermal implant-bioabsorbable gestrinone pellet use in women with pelvic pain secondary to endometriosis after 6 months of Gestrinone pellet insertion versus placebo pellet. PK profile of the gestrinone pellet will be monitored.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind and placebo-controlled study to evaluate the safety and tolerability of of subdermal implant-bioabsorbable gestrinone pellet use in women with pelvic pain secondary to endometriosis. The exploratory aim is to compare the use of a gestrinone pellet with a placebo pellet in the results of participant satisfaction, change in pelvic pain intensity, use of rescue pain medication, quality of life, sexual function, and work activity. PK profile of the gestrinone pellet will be monitored. One hundred patients will be randomized in a 1: 1 ratio. Initially, all the patients will undergo insertion of an intrauterine system of levonorgestrel release (Kyleena) as a contraceptive method. On the same day, after randomization, the subdermal implantation of the gestrinone (85 mg) or placebo pellet will be performed. Visits will occur after 3 and 6 months of the pellet insertion. Primary endpoint is a combination of serious adverse events (SAEs) accumulated within 6 months of pellet insertion and collected through spontaneous reporting and/or clinical findings.

ELIGIBILITY:
Inclusion Criteria

1. Willingness to provide informed consent
2. Woman aged between 18 and 50 years
3. Body weight between 50 ± 5 kg and 90 ± 5 kg
4. Pelvic pain secondary to endometriosis surgically treated with refractory symptoms, independent of pain intensity
5. Deep infiltrative endometriosis documented by biopsies (histopathological examination)
6. Last endometriosis surgery at least 3 months before randomization
7. Not planning to become pregnant within 12 months after the screening visit or be surgically sterilized
8. Absence of changes in the breast (BI-RADS1 and BIRADS-2 classification) documented by an imaging report (mammogram for women aged > 40 years or bilateral breast ultrasound for women aged < 40 years) performed less than 12 months before randomization
9. Agreement not to use other hormones (estrogens, androgens and progestins) in any pharmaceutical form during the study

Exclusion Criteria

1. Chronic severe disorders, including metastatic malignancies, end-stage renal disease with or without dialysis, clinically unstable heart disease, or any other disorder that, in the opinion of the investigator, excludes the participant from the study
2. Suspected or confirmed diagnosis of immunodeficiency based on medical history and/or physical or laboratory examination
3. Other medical or psychiatric conditions, including recent laboratory abnormalities (within the last 12 months) that may increase risks to the study participant or, at the discretion of the investigator, make the participant inappropriate for the study
4. Personal history of thromboembolic events
5. Use anticoagulant medication
6. Contraindication to the use of hormonal contraceptives
7. Suspected or confirmed pregnancy
8. Breastfeeding
9. Current or recurrent pelvic inflammatory disease or other conditions that increase the risk of pelvic infections
10. Postpartum endometritis or septic miscarriage in the last 3 months
11. Abnormal uterine bleeding of unknown etiology
12. Congenital or acquired uterine anomalies, including fibroids (leiomyomas or fibromas) that cause distortion of the uterine cavity
13. Uterine or cervical malignancy
14. Suspected or confirmed diagnosis of estrogen-dependent neoplasm, including breast cancer
15. Cervicitis or vaginitis, including bacterial vaginosis or another uncontrolled lower urinary tract infection
16. Cervical dysplasia
17. Active liver disease or dysfunction
18. Benign or malignant liver tumors
19. Allergy or intolerance to levonorgestrel, gestrinone or any other ingredient or component of the Kyleena® formulation or hormonal pellets
20. Previously inserted intrauterine device or levonorgestrel-releasing intrauterine system that has not been removed
21. History of recent trophoblastic disease and continued high HCG levels
22. Bacterial endocarditis
23. Hyperandrogenism at the time of randomization, defined by: hirsutism: Ferriman-Gallwey score ≥ 8; clitoromegaly: defined by the Clitoral index ≥ 35 mm2, acne: defined by the IGA scale (Investigator's global assessment) grade 5 - severe inflammatory acne dominates the area and there is a large number of comedones, pustules, papules and cystic acne; alopecia with sequelae of scalp thinning
24. Diagnosis of polycystic ovary syndrome
25. Participation in another pharmacotherapeutic or investigational medical device study within 30 days prior to the start of study treatment
26. Tobacco Use
27. Use of testosterone-derived hormones and analogues in the last month

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Combination of serious adverse events (SAEs) accumulated within 6 months of gestrinone or placebo pellet insertion and collected through spontaneous reporting and/or clinical findings | From randomization to the end of study on Day 180
  Proportion of patients who do NOT have SAEs: defined as a combination of death, conditions that threat or present risk to life, conditions needing hospitalization or prolonging the pre-existing hospitalization, conditions causing disability or permanent damage, conditions leading to a congenital anomaly and any other significant medical occurrence that, based on appropriate medical judgment, may harm the participant and/or require medical or surgical intervention to prevent any of the other aforementioned occurrences.

SECONDARY OUTCOMES:
Androgenization | pre-insertion assessment of the pellet (baseline), 3 and 6 months after insertion of the gestrinone or placebo pellet
  Number of participants who experience androgenization defined by: Hirsutism (Ferriman-Gallwey Score ≥ 8), Clitoromegaly (Clitoridian index ≥ 35 mm2), Acne (IGA scale grade 5 - severe inflammatory acne dominates the area and there are large numbers of comedones, pustules, papules, and cystic acne), Alopecia, oiliness of the skin, and deepening of the voice
Plasma concentration of steroid hormones | pre-insertion of the pellet (baseline) and 3 months after pellet insertion of the gestrinone or placebo pellet
  plasma concentration of total testosterone, free testosterone, and SHBG
Lipid profile | pre-insertion of the pellet (baseline) and 3 months after pellet insertion of the gestrinone or placebo pellet
  Serum levels of total cholesterol, HDL-C, VLDL-C, and triglycerides
Uterine Bleeding Pattern | daily for 3 months after pellet insertion of the gestrinone or placebo pellet
  Changes in uterine bleeding pattern (spotting/bleeding)
Hematological disorders | pre-insertion of the pellet (baseline) and 3 months after pellet insertion of the gestrinone or placebo pellet
  Number of participants with decreased lymphocyte count < 500/mm3 (or < 0.5 × 109/l); decrease in neutrophil count < 500/mm3 (or < 0.5 × 109/l); decrease in platelet count < 30,000/mm3 (or < 30.0 × 109/l); and anemia with decreased Hb < 7.0 g/dl (or < 4.35 mmol/l)
Hepatic adverse events | pre-insertion of the pellet (baseline) and 3 months after pellet insertion of the gestrinone or placebo pellet
  Number of participants with increased ALT or AST > 3 times ULN or baseline, alterations in ALP levels suspected hepatocellular or cholestatic hepatotoxicity
Renal adverse events | pre-insertion of the pellet (baseline) and 3 months after pellet insertion of the gestrinone or placebo pellet
  Number of participants with increased serum creatinine ≥ 1.5 times ULN or baseline; clinically significant increase in serum urea

OTHER OUTCOMES:
Overall participant satisfaction | 3 months after pellet insertion of the gestrinone or placebo pellet
  Median of the participant satisfaction scale (ranging from 1 to 5, from very satisfied to very dissatisfied)
Pelvic pain intensity | pre-insertion assessment of the pellet (baseline), 3 and 6 months after insertion of the gestrinone or placebo pellet
  Median of pelvic pain and dysmenorrhea intensity assessed by the VAS visual analogue scale, from 0 to 10 points where 10 points indicates worst pain
Use of pain relief medication | pre-insertion assessment of the pellet (baseline), 3 and 6 months after insertion of the gestrinone or placebo pellet
  Number of participants who used pain relief medication (analgesics and anti-inflammatories)
Patient-reported Quality of Life | pre-insertion assessment of the pellet (baseline), 3 and 6 months after insertion of the gestrinone or placebo pellet
  Number of participants with changes in the 36-Item Short Form Health Survey (SF-36). SF-36 is a patient-reported outcome (PRO) measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health
Endometriosis Health Profile | pre-insertion of the pellet (baseline) and 3 months after pellet insertion of the gestrinone or placebo pellet
  Number of participants with changes in the Endometriosis Health Profile Questionnaire (EHP-30). The Endometriosis Health Profile Questionnaire is a Health Related Quality of Life (HRQoL) patient self-report PRO, used to measure the wide range of effects that endometriosis can have on women's lives: pain, control and powerlessness, social support, emotional well-being, and self-image, range from 0-100, higher values indicate worse health status
Serum total gestrinone concentration | pre-insertion of the pellet (baseline) and 24 hours; 7 days, 14 days , 21 days , 28 days , 56 days, 84 days, 112 days, 140 days and 168 days post-insertion
  Multiple blood sample will be collected before pellet implantation and 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Area under the curve (AUC(0 ∞)) | pre-insertion of the pellet (baseline) and 24 hours; 7 days, 14 days , 21 days , 28 days , 56 days, 84 days, 112 days, 140 days and 168 days post-insertion
  Multiple blood sample will be collected before pellet implantation and 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Maximum concentration (Cmax) | pre-insertion of the pellet (baseline) and 24 hours; 7 days, 14 days , 21 days , 28 days , 56 days, 84 days, 112 days, 140 days and 168 days post-insertion
  Multiple blood sample will be collected before pellet implantation and 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Time to reach maximum concentration (tmax) | pre-insertion of the pellet (baseline) and 24 hours; 7 days, 14 days , 21 days , 28 days , 56 days, 84 days, 112 days, 140 days and 168 days post-insertion
  Multiple blood sample will be collected before pellet implantation and 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Half Life (t1/2) | pre-insertion of the pellet (baseline) and 24 hours; 7 days, 14 days , 21 days , 28 days , 56 days, 84 days, 112 days, 140 days and 168 days post-insertion
  Multiple blood sample will be collected before pellet implantation and 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ramacciotti, MD, PhD, Study Chair — Science Valley Research Institute; André Luiz M Oliveira, MD, MHS, Principal Investigator — Science Valley Research Institute
Locations (1):
- Science Valley Research Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Becker CM, Bokor A, Heikinheimo O, Horne A, Jansen F, Kiesel L, King K, Kvaskoff M, Nap A, Petersen K, Saridogan E, Tomassetti C, van Hanegem N, Vulliemoz N, Vermeulen N; ESHRE Endometriosis Guideline Group. ESHRE guideline: endometriosis. Hum Reprod Open. 2022 Feb 26;2022(2):hoac009. doi: 10.1093/hropen/hoac009. eCollection 2022. PMID 35350465
- [Background] Coutinho EM. Treatment of endometriosis with gestrinone (R-2323), a synthetic antiestrogen, antiprogesterone. Am J Obstet Gynecol. 1982 Dec 15;144(8):895-8. doi: 10.1016/0002-9378(82)90180-6. PMID 6216812
- [Background] Venturini PL, Bertolini S, Brunenghi MC, Daga A, Fasce V, Marcenaro A, Cimato M, De Cecco L. Endocrine, metabolic, and clinical effects of gestrinone in women with endometriosis. Fertil Steril. 1989 Oct;52(4):589-95. doi: 10.1016/s0015-0282(16)60969-x. PMID 2806598
- [Background] Gestrinone versus a gonadotropin-releasing hormone agonist for the treatment of pelvic pain associated with endometriosis: a multicenter, randomized, double-blind study. Gestrinone Italian Study Group. Fertil Steril. 1996 Dec;66(6):911-9. doi: 10.1016/s0015-0282(16)58682-8. PMID 8941054
- [Background] Devogelaer JP, Nagant de Deuxchaisnes C, Donnez J. Endometriosis. Lancet. 1993 Jan 30;341(8840):312-3. doi: 10.1016/0140-6736(93)92673-h. No abstract available. PMID 8093956
- [Background] Malavasi A, Ribeiro CM, Agati LB, Silva Filho A, Berger C, Schor E, Comin A, Bezerra Neto EJ, Oliveira TH, Caldas PR, Lopes F, Westphalen N, Vieira F, Socca EAR, Komar D, Ramacciotti E. Rationale and design of the GLADE study: a randomized, multicenter, double-blind, placebo-controlled trial evaluating the safety and efficacy of gestrinone subdermal bioabsorbable pellet in endometriosis-related pelvic pain. Ann Med. 2025 Dec;57(1):2527352. doi: 10.1080/07853890.2025.2527352. Epub 2025 Jul 11. PMID 40641309